CLINICAL TRIAL: NCT01080209
Title: Safety Extension Study to Evaluate the Biodegradation of the Brimonidine Tartrate Posterior Segment Drug Delivery System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single
Other Study IDs: 190342-033D
Record Dates: First submitted 2010-02-26; First posted 2010-03-04 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Patients Who Participated in an Intravitreal Brimo PS DDS® Study
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- Brimo PS DDS® 400 μg (2 implants) (Experimental): Patients who received Brimo PS DDS® 400 μg (2 implants) in a previous study.
  Interventions: Drug: Brimo PS DDS®
- Brimo PS DDS® 400 μg (1 implant) (Experimental): Patients who received Brimo PS DDS® 400 μg (1 implant) in a previous study.
  Interventions: Drug: Brimo PS DDS®
- Brimo PS DDS® 200 μg (2 implants) (Experimental): Patients who received Brimo PS DDS® 200 μg (2 implants) in a previous study.
  Interventions: Drug: Brimo PS DDS®
- Brimo PS DDS® 200 μg (1 implant) (Experimental): Patients who received Brimo PS DDS® 200 μg (1 implant) in a previous study.
  Interventions: Drug: Brimo PS DDS®
- Brimo PS DDS® 100 μg (1 implant) (Experimental): Patients who received Brimo PS DDS® 100 μg (1 implant) in a previous study.
  Interventions: Drug: Brimo PS DDS®
- Brimo PS DDS® 50 μg (1 implant) (Experimental): Patients who received Brimo PS DDS® 50 μg (1 implant) in a previous study.
  Interventions: Drug: Brimo PS DDS®
- Sham (Sham Comparator): Patients who received sham in a previous study.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Brimo PS DDS® — Patients who received Brimo PS DDS® intravitreal implant in a previous study.
  Arms: Brimo PS DDS® 100 μg (1 implant); Brimo PS DDS® 200 μg (1 implant); Brimo PS DDS® 200 μg (2 implants); Brimo PS DDS® 400 μg (1 implant); Brimo PS DDS® 400 μg (2 implants); Brimo PS DDS® 50 μg (1 implant)
Other: Sham — Patients who recieved sham in a previous study.
  Arms: Sham

SUMMARY:
This study will evaluate the biodegradation of the brimonidine tartrate posterior segment drug delivery system.

ELIGIBILITY:
Inclusion Criteria:

* Received the most recent sham or active study treatment of intravitreal Brimo PS DDS® no later than 36 months prior to entry into this study and have either completed their previous study, or have exited early from their previous study for any reason
* Applicable studies: Previous Allergan intravitreal Brimo PS DDS® treatment studies

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2010-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (13):
- Artesia, California, United States
- Australia (2):
  - Sydney, New South Wales
  - Westmead, New South Wales
- Brno, Czechia
- Paris, France
- Karlsruhe, Germany
- New Delhi, New Delhi, India
- Tel Aviv, Israel
- Udine, Italy
- Makati, Philippines
- Coimbra, Portugal
- Seoul, South Korea
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients enrolled in this extension study from the following parent studies: 190342-027D, 190342-028D, 190342-030D, 190342-031D, 190342-032D, and 190342-036. No treatment was administered in this study, so the treatment groups reflect the treatments received in the parent studies.
Period: Overall Study
Arm/Group | Brimo PS DDS® 400 μg (2 Implants) | Brimo PS DDS® 400 μg (1 Implant) | Brimo PS DDS® 200 μg (2 Implants) | Brimo PS DDS® 200 μg (1 Implant) | Brimo PS DDS® 100 μg (1 Implant) | Brimo PS DDS® 50 μg (1 Implant) | Sham
Started | 28 | 53 | 33 | 42 | 6 | 2 | 51
Completed | 22 | 42 | 28 | 37 | 6 | 2 | 44
Not Completed | 6 | 11 | 5 | 5 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brimo PS DDS® 400 μg (2 Implants) | Brimo PS DDS® 400 μg (1 Implant) | Brimo PS DDS® 200 μg (2 Implants) | Brimo PS DDS® 200 μg (1 Implant) | Brimo PS DDS® 100 μg (1 Implant) | Brimo PS DDS® 50 μg (1 Implant) | Sham | Total
Number analyzed (Participants) | 28 | 53 | 33 | 42 | 6 | 2 | 51 | 215
Age, Customized [Number; unit: Participants]
  18 to 64 years | 2 | 23 | 3 | 20 | 3 | 0 | 20 | 71
  Between 65 and 84 years | 19 | 29 | 24 | 19 | 3 | 1 | 26 | 121
  ≥85 years | 7 | 1 | 6 | 3 | 0 | 1 | 5 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 17 | 20 | 3 | 2 | 21 | 106
  Male | 9 | 29 | 16 | 22 | 3 | 0 | 30 | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With No Visible Implants in the Study Eye
Description: Implants administered during the parent study are evaluated during this study to determine if they have completely degraded. The time frame is evaluated from the point of the first treatment in the parent study.
Time Frame: Month 36
Population: Safety Population: all enrolled patients, who received a sham or active study treatment of intravitreal Brimonidine Tartrate PS DDS in the parent study
Measure: Number; unit: Patients
Arm/Group | Brimo PS DDS® 400 μg (2 Implants) | Brimo PS DDS® 400 μg (1 Implant) | Brimo PS DDS® 200 μg (2 Implants) | Brimo PS DDS® 200 μg (1 Implant) | Brimo PS DDS® 100 μg (1 Implant) | Brimo PS DDS® 50 μg (1 Implant) | Sham
Number analyzed (Participants) | 23 | 42 | 30 | 37 | 6 | 2 | 46
Patients | 14 | 37 | 26 | 35 | 6 | 2 | 46

2. Secondary Outcome: Number of Patients With Vision Loss in the Study Eye
Description: Vision loss is assessed by Best Corrected Visual Acuity (BCVA) in the study eye. BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). Severe vision loss is a ≥30 letter decrease in BCVA. Moderate vision loss is a ≥15 and <30 letter decrease in BCVA. No or mild vision loss is <15 letter decrease in BCVA. Baseline of the parent study is defined as the point of the first study treatment.
Time Frame: Baseline of Parent Study, Month 36
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Brimo PS DDS® 400 μg (2 Implants) | Brimo PS DDS® 400 μg (1 Implant) | Brimo PS DDS® 200 μg (2 Implants) | Brimo PS DDS® 200 μg (1 Implant) | Brimo PS DDS® 100 μg (1 Implant) | Brimo PS DDS® 50 μg (1 Implant) | Sham
Number analyzed (Participants) | 23 | 42 | 30 | 37 | 6 | 2 | 46
Patients
  Severe Vision Loss | 3 | 1 | 1 | 0 | 0 | 0 | 4
  Moderate Vision Loss | 6 | 0 | 6 | 1 | 0 | 0 | 6
  No or Mild Vision Loss | 14 | 41 | 23 | 36 | 6 | 2 | 36

ADVERSE EVENTS:
Arm/Group | Brimo PS DDS® 400 μg (2 Implants) | Brimo PS DDS® 400 μg (1 Implant) | Brimo PS DDS® 200 μg (2 Implants) | Brimo PS DDS® 200 μg (1 Implant) | Brimo PS DDS® 100 μg (1 Implant) | Brimo PS DDS® 50 μg (1 Implant) | Sham
Serious Adverse Events (participants affected / at risk) | 8/28 | 11/53 | 7/33 | 7/42 | 2/6 | 0/2 | 16/51
Other Adverse Events (participants affected / at risk) | 13/28 | 30/53 | 17/33 | 25/42 | 4/6 | 2/2 | 26/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Brimo PS DDS® 400 μg (2 Implants) (N=28) | Brimo PS DDS® 400 μg (1 Implant) (N=53) | Brimo PS DDS® 200 μg (2 Implants) (N=33) | Brimo PS DDS® 200 μg (1 Implant) (N=42) | Brimo PS DDS® 100 μg (1 Implant) (N=6) | Brimo PS DDS® 50 μg (1 Implant) (N=2) | Sham (N=51)
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1/19 | 0/24 | 0/17 | 1/20 | 0/3 | 0 | 0/21
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Age-Related Macular Degeneration (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 1/19 | 0/24 | 0/17 | 0/20 | 0/3 | 0 | 0/21
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterocele (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 1/19 | 0/24 | 0/17 | 0/20 | 0/3 | 0 | 0/21
Sudden Cardiac Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual Acuity Reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal Detachment (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory Arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0/9 | 1/29 | 0/16 | 0/22 | 0/3 | 0/0 | 0/30
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinal Vein Occlusion (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Anterior Chamber Inflammation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Open Angle Glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral Artery Stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral Vascular Disorder (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9 | 0/29 | 0/16 | 1/22 | 0/3 | 0/0 | 0/30
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9 | 0/29 | 0/16 | 0/22 | 1/3 | 0/0 | 0/30
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intermittent Claudication (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Jaw Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis Ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pubis Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Optic Atrophy (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhagic Stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Brimo PS DDS® 400 μg (2 Implants) (N=28) | Brimo PS DDS® 400 μg (1 Implant) (N=53) | Brimo PS DDS® 200 μg (2 Implants) (N=33) | Brimo PS DDS® 200 μg (1 Implant) (N=42) | Brimo PS DDS® 100 μg (1 Implant) (N=6) | Brimo PS DDS® 50 μg (1 Implant) (N=2) | Sham (N=51)
Cataract (Eye disorders) | 3 | 6 | 0 | 6 | 0 | 0 | 6
Visual Acuity Reduced (Eye disorders) | 3 | 3 | 3 | 5 | 0 | 0 | 0
Age-Related Macular Degeneration (Eye disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 0
Vitreous Detachment (Eye disorders) | 2 | 0 | 2 | 4 | 0 | 0 | 4
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 3
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous Floaters (Eye disorders) | 0 | 5 | 3 | 3 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3 | 0 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal Haemorrhage (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Posterior Capsule Opacification (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4
Intraocular Pressure Increased (Investigations) | 0 | 6 | 0 | 4 | 0 | 0 | 4
Dry Eye (Eye disorders) | 0 | 5 | 2 | 4 | 0 | 0 | 0
Macular Fibrosis (Eye disorders) | 0 | 4 | 0 | 3 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 3 | 3 | 4 | 0 | 0 | 4
Optic Disc Haemorrhage (Eye disorders) | 0 | 3 | 2 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 3 | 0 | 4 | 0 | 0 | 5
Macular Degeneration (Eye disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0/9 | 0/29 | 0/16 | 3/22 | 0/3 | 0/0 | 0/30
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Glare (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cataract Cortical (Eye disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis Media Chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Restless Legs Syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stress Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract Subscapular (Eye disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.